CLINICAL TRIAL: NCT03956901
Title: Peroperative and Postoperative Effects of Goal Directed Fluid Therapy in Gynecological Staging Surgery
Brief Title: Goal Directed Fluid Management , Pvi
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Responsible Party: Principal Investigator, Güneş Özlem Yıldız, principal investigator, Bakirkoy Dr. Sadi Konuk Research and Training Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2019/152
Record Dates: First submitted 2019-05-17; First posted 2019-05-21 (Actual); Last update posted 2020-07-13 (Actual); Status verified 2020-05

CONDITIONS: Fluid Overload
MeSH Terms: conditions — Edema

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Liberal Fluid Management (Experimental): liberal fluid management: 500 ml bolus crystalloid after 4-8 ml/kg/h infusion during surgery total amount of crystalloid volume of fluid infused during gycnecologcy l surgery fluid infused during whole procedure 4-8 ml/kg/h infusion during surgery If MAP <65 mmHg or <30%of basal value, infuse 250 ml cyristaloid/Gelofusine bolus and 5 mcg efedrin If MAP>65 mmHg no intervention
  Interventions: Other: pvi guided fluid management
- pvi guided fluid management (Experimental): GDFM Group: 500 ml bolus crystalloid after
  2 ml \ kg crystalloid infusion to be started
  If PVI <13 MAP is <65 mmHg, continue infusion of fluid, 1-2 µg NE bolus to be entered after 5 min.
  PVI <13 MAP> 65 mmHg to continue fluid infusion If PVI> 13 MAP <65 mmHg, 250 ml bolus crystalloid \ colloid will be given and bolus 1-2 µg NE, If it continues after 5 minutes, liquid and NE doses will be repeated. Liquid treatment will be continued until PVI <13.
  PVI> 13 MAP <65 mmHg 250 ml bolus fluid to be given, if continued 5 minutes later to be repeated,repetition of fluid will continue until PVl <13.
  Interventions: Other: pvi guided fluid management

INTERVENTIONS:
Other: pvi guided fluid management — GDFM Group: 500 ml bolus crystalloid after
  2 ml \ kg crystalloid infusion to be started
  If PVI <13 MAP is <65 mmHg, continue infusion of fluid, 1-2 µg NE bolus to be entered after 5 min.
  PVI <13 MAP> 65 mmHg to continue fluid infusion If PVI> 13 MAP <65 mmHg, 250 ml bolus crystalloid \ colloid will be given and bolus 1-2 µg NE, If it continues after 5 minutes, liquid and NE doses will be repeated. Liquid treatment will be continued until PVI <13.
  PVI> 13 MAP <65 mmHg 250 ml bolus fluid to be given, if continued 5 minutes later to be repeated,repetition of fluid will continue until PVl <13.
  Other Names: liberal guided

SUMMARY:
The first objective of this study is to compare the liberal fluid management (LFM) with PVI guided goal-directed fluid management (GDFM) in gynecologic oncologic cases in terms of controlled intraoperative fluid balance, blood lactate levels, hemodynamic parameters, and postoperative serum creatinine levels. 112 patients who are in ASA I-II-lll risk groups included in this prospective study.

DETAILED DESCRIPTION:
Objectives: The first objective of the investigators's study was to compare the liberal fluid management (LFM) with PVI guided goal-directed fluid management (GDFM) in terms of controlled intraoperative fluid volume, surgical end-point fluid balance, blood lactate and serum creatinine levels.

The investigators's secondary purpose was to compare the effects of different fluid regimens on the postoperative kidney injury and the duration of hospital stay.

Methods: The study included 112 American Society of Anesthesiologists (ASA) grade I ,ll and lll patients, aged above 18 and undergoing elective gynecologic oncologic case . After premedication with 0.03 mg /kg i.v. midazolam, all patients were started an i.v. infusion of 500 mL 0.9 % NaCl until the end of anesthesia induction.

After the anesthesia induction, while 0.9 % NaCl at rate of 2 mL/kg/h was infused in PVI- guided GDFM group, a 250-mL bolus cyristalloid/kolloid injection was administered when PVI was higher than 13 % over 5 min. While 0.9 % NaCl at rate of 4- 8 mL/kg/h was infused in LFM group, a 250-ml bolus cyristalloid/ kolloid injection was administered when the mean arterial blood pressure (MAP) decreased below 65 mmHg. In both groups, when MAP was still < 65 mmHg after fluid bolus infusion, 5 mg i.v. bolus ephedrine was administered. The data collected during intraoperative period, such as heart rate, MAP, arterial blood gas samples (Ph, arterial oxygen pressure (PaO2), arterial carbon dioxide pressure (PaCO2), HCO3 level, hemoglobin, blood lactate level) were recorded. Hemoglobin, Na, K, Cl, serum creatinine, blood lactate and serum albumin scores were measured preoperatively, and up to 24 hours postoperative.

In the first 24 hours after surgery, urine output, need for blood transfusion ,lokositoz,fever,stay in icu and length of hospital stay were recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Gynecological oncologic cases
2. Patients over 18 years old
3. ASA 1-2-3 patients

Exclusion Criteria:

1. Patients with peripheral arterial disease
2. Patients with non-sinus rhythm, arrhythmia, atrial fibrillation
3. Patients with entry MAP <65 mmHg
4. Patients with advanced renal and hepatic impairment
5. Mental retarded and non-cooperative patients
6. Patients with advanced heart failure, EF <30%
7. Patients have massive bleeding in the perioperative period, need for massive transfusion
8. Patients have acute pulmonary pathology
9. Patients with anaphylaxis who developed a blood product reaction
10. Patients who do not allow a tidal volume of 8ml / kg in a mechanical ventilator

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2019-04-08 (Actual); Primary Completion 2019-05-08 (Actual); Study Completion 2020-06-20 (Actual)

PRIMARY OUTCOMES:
fluid management | 3-4 hours
  total fluid given durin operation

CONTACTS AND LOCATIONS:
Overall Officials: güneş özlem yildiz, Principal Investigator — bakırköy Dr. Sadi Konuk Education hospital
Locations (1):
- Bakırköy Dr sadi konuk Education hospital, Istanbul, Turkey (Türkiye)